CLINICAL TRIAL: NCT02381457
Title: SNP-based Microdeletion and Aneuploidy RegisTry
Brief Title: SNP-based Microdeletion and Aneuploidy RegisTry (SMART)
Acronym: SMART
Status: Completed | Type: Observational
Sponsor: Natera, Inc. (Industry)
Collaborators: George Washington University (Other); University of California, San Francisco (Other); Montefiore Medical Center (Other); Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 14-024-NPT
Record Dates: First submitted 2015-03-02; First posted 2015-03-06 (Estimated); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: 22q11 Deletion Syndrome; DiGeorge Syndrome; Trisomy 21; Trisomy 18; Trisomy 13; Monosomy X; Sex Chromosome Abnormalities; Cri-du-Chat Syndrome; Angelman Syndrome; Prader-Willi Syndrome; 1p36 Deletion Syndrome
Keywords: Microdeletion Syndrome; Aneuploidy; 22q; Non-Invasive Prenatal Screening; DiGeorge Syndrome
MeSH Terms: conditions — 22q11 Deletion Syndrome; DiGeorge Syndrome; Down Syndrome; Trisomy 18 Syndrome; Trisomy 13 Syndrome; Turner Syndrome; Sex Chromosome Aberrations; Cri-du-Chat Syndrome; Angelman Syndrome; Prader-Willi Syndrome; Chromosome 1p36 Deletion Syndrome; Aneuploidy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — * Maternal residual blood sample
  * Placental tissue
  * Child dried blood spot
  * Child buccal sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnancies undergoing prenatal microdeletion screening: Pregnant women undergoing non-invasive prenatal screening for microdeletion and aneuploidy syndromes.
  No drug will be administrated, this cohort will undergo a non invasive prenatal blood test and then follow up data and specimens will be collected for research analysis.

SUMMARY:
This multi-center prospective observational study is designed to track birth outcomes and perinatal correlates to the Panorama prenatal screening test in the general population among ten thousand women who present clinically and elect Panorama microdeletion and aneuploidy screening as part of their routine care. The primary objective is to evaluate the performance of Single Nucleotide Polymorphism (SNP)-based Non Invasive Prenatal Testing (NIPT) for 22q11.2 microdeletion (DiGeorge syndrome) in this large cohort of pregnant women. This will be done by performing a review of perinatal medical records and obtaining biospecimens after birth to perform genetic diagnostic testing for 22q11.2 deletion. Results from the follow-up specimens will be compared to those obtained by the Panorama screening test to determine test performance. Specific test performance parameters will include: PPV, specificity, and sensitivity.

DETAILED DESCRIPTION:
The primary objective is to determine in a prospective study the performance of SNP based NIPT for the 22q11.2 microdeletion (DiGeorge syndrome) in a large cohort of pregnant women clinically opting for this form of screening. Specific test performance parameters will include: positive predictive value (PPV), specificity, and sensitivity.

Secondary objectives include:

1. Determine the test performance (PPV, specificity) of SNP based NIPT for detecting other microdeletion syndromes available in the Panorama microdeletion panel (e.g., 1p36 deletion, Cri-du-chat, Prader-Willi, and Angelman) individually and all combined (including 22q11.2). Given the incidences of <1:5000, the confidence intervals are expected to be large.
2. Determine the failure ('no call') rate for the Next-generation Aneuploidy Test Using SNPs (NATUS) method for 22q11.2 detection, as well as for aneuploidy.
3. Determine whether a more precise risk for aneuploidy can be generated in the setting of low fetal fraction by incorporating maternal BMI (adjusted fetal fraction percentile).
4. Assess whether low fetal fraction is associated with specific ultrasound findings that may indicate aneuploidy (e.g. triploidy, trisomy 13 and 18).
5. Investigate the relationship between NIPT and sonographic (nuchal translucency and anatomy survey) markers and serum markers from 1st and 2nd trimester aneuploidy screening.
6. Determine sensitivity, specificity, and PPV for chromosomal aneuploidies and sex chromosome abnormalities.
7. Perform detailed assessment of false positive aneuploidy samples to better understand sources of error, including placental studies to further refine issues surrounding mosaicism as NIPT represents circulating placental DNA.
8. Investigate any relationships between circulating placental DNA (fetal fraction) or other test parameters including potential genotypic markers, and outcomes related to abnormal placentation (including but not limited to preeclampsia, small for gestational age and morbidly adherent placenta).
9. Investigate other risk factors that may impact risk assessment for microdeletions including sonographic findings consistent with 22q11.2 (cardiac anomalies and thymus size).

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Receiving Panorama prenatal screening test for both microdeletions (at least 22q11.2) and aneuploidy
* Planned hospital delivery
* Gestational age of ≥ 9 weeks, 0 days based on clinical information and evaluation.
* Able to provide informed consent

Exclusion Criteria:

* Received results of the Panorama test prior to enrollment
* Organ transplant recipient
* Egg donor used

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 20960 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
22q11.2 Snp-based non-invasive prenatal screening test performance, including positive predictive value (PPV), specificity, and sensitivity | 3 years
  To determine in a prospective study the performance of SNP based NIPT for the 22q11.2 microdeletion (DiGeorge syndrome) in a large cohort of pregnant women clinically opting for this form of screening.

SECONDARY OUTCOMES:
Combined microdeletion syndrome screening test performance | 3 years
  Determine the test performance (PPV, specificity) of SNP based NIPT for detecting other microdeletion syndromes available in the Panorama microdeletion panel (e.g., 1p36 deletion, Cri-du-chat, Prader-Willi, and Angelman) individually and all combined (including 22q11.2). Given the incidences of <1:5000, the confidence intervals are expected to be large.
No call rate | 3 years
  Determine the failure ('no call') rate for the NATUS method for 22q11.2 detection, as well as for aneuploidy.
Low fetal fraction aneuploidy risk refinement | 3 years
  Determine whether a more precise risk for aneuploidy can be generated in the setting of low fetal fraction by incorporating maternal BMI (adjusted fetal fraction percentile), or whether low fetal fraction is associated with specific ultrasound findings that may indicate aneuploidy (e.g. triploidy, trisomy 13 and 18).
Placental mosaicism exploration | 3 years
  Perform detailed assessment of false positive aneuploidy samples to better understand sources of error, including placental studies to further refine issues surrounding mosaicism as NIPT represents circulating placental DNA.
Placental complications exploration | 3 years
  Investigate any relationships between circulating placental DNA (fetal fraction) or other test parameters including potential genotypic markers, and outcomes related to abnormal placentation (including but not limited to preeclampsia, small for gestational age and morbidly adherent placenta).

CONTACTS AND LOCATIONS:
Overall Officials: Peer Dar, MD, Principal Investigator — Montefiore Medical Center; Mary Norton, MD, Principal Investigator — University of California, San Francisco
Locations (21):
- United States (16):
  - University of California, San Francisco, San Francisco, California
  - Cooper University Hospital, Camden, New Jersey
  - Virtua, Mount Laurel, New Jersey
  - St. Peter's University, New Brunswick, New Jersey
  - Complete Women's Healthcare, Garden City, New York
  - North Shore University Hospital, Manhasset, New York
  - Madonna Perinatal, Mineola, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - New York University, New York, New York
  - Icahn School of Medicine Mt Sinai, New York, New York
  - Columbia University, New York, New York
  - Montefiore Medical Center, New York, New York
  - Suffolk OB, Port Jefferson, New York
  - North Austin Maternal Fetal Medicine, Austin, Texas
  - Zeid Women's Health Center, Longview, Texas
  - University of Utah, Salt Lake City, Utah
- Royal Prince Alfred, Camperdown, New South Wales, Australia
- Royal College Surgeons in Ireland, Dublin, Ireland
- Dexeus, Barcelona, Spain
- Sahlgrenska University Hospital, Gothenburg, Sweden
- St. George University Hospital, London, United Kingdom

REFERENCES:
- [Background] American College of Obstetricians and Gynecologists Committee on Genetics. Committee Opinion No. 581: the use of chromosomal microarray analysis in prenatal diagnosis. Obstet Gynecol. 2013 Dec;122(6):1374-7. doi: 10.1097/01.AOG.0000438962.16108.d1. PMID 24264715
- [Result] Pergament E, Cuckle H, Zimmermann B, Banjevic M, Sigurjonsson S, Ryan A, Hall MP, Dodd M, Lacroute P, Stosic M, Chopra N, Hunkapiller N, Prosen DE, McAdoo S, Demko Z, Siddiqui A, Hill M, Rabinowitz M. Single-nucleotide polymorphism-based noninvasive prenatal screening in a high-risk and low-risk cohort. Obstet Gynecol. 2014 Aug;124(2 Pt 1):210-218. doi: 10.1097/AOG.0000000000000363. PMID 25004354
- [Result] Ehrich M, Deciu C, Zwiefelhofer T, Tynan JA, Cagasan L, Tim R, Lu V, McCullough R, McCarthy E, Nygren AO, Dean J, Tang L, Hutchison D, Lu T, Wang H, Angkachatchai V, Oeth P, Cantor CR, Bombard A, van den Boom D. Noninvasive detection of fetal trisomy 21 by sequencing of DNA in maternal blood: a study in a clinical setting. Am J Obstet Gynecol. 2011 Mar;204(3):205.e1-11. doi: 10.1016/j.ajog.2010.12.060. Epub 2011 Feb 18. PMID 21310373
- [Result] Palomaki GE, Kloza EM, Lambert-Messerlian GM, Haddow JE, Neveux LM, Ehrich M, van den Boom D, Bombard AT, Deciu C, Grody WW, Nelson SF, Canick JA. DNA sequencing of maternal plasma to detect Down syndrome: an international clinical validation study. Genet Med. 2011 Nov;13(11):913-20. doi: 10.1097/GIM.0b013e3182368a0e. PMID 22005709
- [Result] Sehnert AJ, Rhees B, Comstock D, de Feo E, Heilek G, Burke J, Rava RP. Optimal detection of fetal chromosomal abnormalities by massively parallel DNA sequencing of cell-free fetal DNA from maternal blood. Clin Chem. 2011 Jul;57(7):1042-9. doi: 10.1373/clinchem.2011.165910. Epub 2011 Apr 25. PMID 21519036
- [Result] Benn P, Cuckle H, Pergament E. Genome-wide fetal aneuploidy detection by maternal plasma DNA sequencing. Obstet Gynecol. 2012 Jun;119(6):1270; author reply 1270-1. doi: 10.1097/AOG.0b013e318258c401. No abstract available. PMID 22617594
- [Result] Palomaki GE, Deciu C, Kloza EM, Lambert-Messerlian GM, Haddow JE, Neveux LM, Ehrich M, van den Boom D, Bombard AT, Grody WW, Nelson SF, Canick JA. DNA sequencing of maternal plasma reliably identifies trisomy 18 and trisomy 13 as well as Down syndrome: an international collaborative study. Genet Med. 2012 Mar;14(3):296-305. doi: 10.1038/gim.2011.73. Epub 2012 Feb 2. PMID 22281937
- [Result] Sparks AB, Struble CA, Wang ET, Song K, Oliphant A. Noninvasive prenatal detection and selective analysis of cell-free DNA obtained from maternal blood: evaluation for trisomy 21 and trisomy 18. Am J Obstet Gynecol. 2012 Apr;206(4):319.e1-9. doi: 10.1016/j.ajog.2012.01.030. Epub 2012 Jan 26. PMID 22464072
- [Result] Norton ME, Brar H, Weiss J, Karimi A, Laurent LC, Caughey AB, Rodriguez MH, Williams J 3rd, Mitchell ME, Adair CD, Lee H, Jacobsson B, Tomlinson MW, Oepkes D, Hollemon D, Sparks AB, Oliphant A, Song K. Non-Invasive Chromosomal Evaluation (NICE) Study: results of a multicenter prospective cohort study for detection of fetal trisomy 21 and trisomy 18. Am J Obstet Gynecol. 2012 Aug;207(2):137.e1-8. doi: 10.1016/j.ajog.2012.05.021. Epub 2012 Jun 1. PMID 22742782
- [Result] Nicolaides KH, Syngelaki A, Gil M, Atanasova V, Markova D. Validation of targeted sequencing of single-nucleotide polymorphisms for non-invasive prenatal detection of aneuploidy of chromosomes 13, 18, 21, X, and Y. Prenat Diagn. 2013 Jun;33(6):575-9. doi: 10.1002/pd.4103. Epub 2013 Apr 24. PMID 23613152
- [Result] Nicolaides KH, Syngelaki A, del Mar Gil M, Quezada MS, Zinevich Y. Prenatal detection of fetal triploidy from cell-free DNA testing in maternal blood. Fetal Diagn Ther. 2014;35(3):212-7. doi: 10.1159/000355655. Epub 2013 Oct 10. PMID 24135152
- [Result] Samango-Sprouse C, Banjevic M, Ryan A, Sigurjonsson S, Zimmermann B, Hill M, Hall MP, Westemeyer M, Saucier J, Demko Z, Rabinowitz M. SNP-based non-invasive prenatal testing detects sex chromosome aneuploidies with high accuracy. Prenat Diagn. 2013 Jul;33(7):643-9. doi: 10.1002/pd.4159. Epub 2013 Jun 20. PMID 23712453
- [Result] Wapner RJ, Martin CL, Levy B, Ballif BC, Eng CM, Zachary JM, Savage M, Platt LD, Saltzman D, Grobman WA, Klugman S, Scholl T, Simpson JL, McCall K, Aggarwal VS, Bunke B, Nahum O, Patel A, Lamb AN, Thom EA, Beaudet AL, Ledbetter DH, Shaffer LG, Jackson L. Chromosomal microarray versus karyotyping for prenatal diagnosis. N Engl J Med. 2012 Dec 6;367(23):2175-84. doi: 10.1056/NEJMoa1203382. PMID 23215555
- [Result] Wapner RJ, Babiarz JE, Levy B, Stosic M, Zimmermann B, Sigurjonsson S, Wayham N, Ryan A, Banjevic M, Lacroute P, Hu J, Hall MP, Demko Z, Siddiqui A, Rabinowitz M, Gross SJ, Hill M, Benn P. Expanding the scope of noninvasive prenatal testing: detection of fetal microdeletion syndromes. Am J Obstet Gynecol. 2015 Mar;212(3):332.e1-9. doi: 10.1016/j.ajog.2014.11.041. Epub 2014 Dec 2. PMID 25479548
- [Result] Vora NL, O'Brien BM. Noninvasive prenatal testing for microdeletion syndromes and expanded trisomies: proceed with caution. Obstet Gynecol. 2014 May;123(5):1097-1099. doi: 10.1097/AOG.0000000000000237. PMID 24785862
- [Result] Taglauer ES, Wilkins-Haug L, Bianchi DW. Review: cell-free fetal DNA in the maternal circulation as an indication of placental health and disease. Placenta. 2014 Feb;35 Suppl(Suppl):S64-8. doi: 10.1016/j.placenta.2013.11.014. Epub 2013 Dec 1. PMID 24388429
- [Result] Knight M, Redman CW, Linton EA, Sargent IL. Shedding of syncytiotrophoblast microvilli into the maternal circulation in pre-eclamptic pregnancies. Br J Obstet Gynaecol. 1998 Jun;105(6):632-40. doi: 10.1111/j.1471-0528.1998.tb10178.x. PMID 9647154
- [Result] Dar P, Curnow KJ, Gross SJ, Hall MP, Stosic M, Demko Z, Zimmermann B, Hill M, Sigurjonsson S, Ryan A, Banjevic M, Kolacki PL, Koch SW, Strom CM, Rabinowitz M, Benn P. Clinical experience and follow-up with large scale single-nucleotide polymorphism-based noninvasive prenatal aneuploidy testing. Am J Obstet Gynecol. 2014 Nov;211(5):527.e1-527.e17. doi: 10.1016/j.ajog.2014.08.006. Epub 2014 Aug 8. PMID 25111587
- [Result] Amos-Landgraf JM, Ji Y, Gottlieb W, Depinet T, Wandstrat AE, Cassidy SB, Driscoll DJ, Rogan PK, Schwartz S, Nicholls RD. Chromosome breakage in the Prader-Willi and Angelman syndromes involves recombination between large, transcribed repeats at proximal and distal breakpoints. Am J Hum Genet. 1999 Aug;65(2):370-86. doi: 10.1086/302510. PMID 10417280
- [Result] Roberts JM, Myatt L, Spong CY, Thom EA, Hauth JC, Leveno KJ, Pearson GD, Wapner RJ, Varner MW, Thorp JM Jr, Mercer BM, Peaceman AM, Ramin SM, Carpenter MW, Samuels P, Sciscione A, Harper M, Smith WJ, Saade G, Sorokin Y, Anderson GB; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Vitamins C and E to prevent complications of pregnancy-associated hypertension. N Engl J Med. 2010 Apr 8;362(14):1282-91. doi: 10.1056/NEJMoa0908056. PMID 20375405
- [Result] Tranquilli AL, Emanuelli M. The thrombophilic fetus. Med Hypotheses. 2006;67(5):1226-9. doi: 10.1016/j.mehy.2006.04.046. Epub 2006 Jul 11. PMID 16814942
- [Result] Faiz AS, Ananth CV. Etiology and risk factors for placenta previa: an overview and meta-analysis of observational studies. J Matern Fetal Neonatal Med. 2003 Mar;13(3):175-90. doi: 10.1080/jmf.13.3.175.190. PMID 12820840
- [Derived] Norton ME, MacPherson C, Demko Z, Egbert M, Malone F, Wapner RJ, Roman AS, Khalil A, Faro R, Madankumar R, Strong N, Haeri S, Silver R, Vohra N, Hyett J, Martin K, Rabinowitz M, Jacobsson B, Dar P. Obstetrical, perinatal, and genetic outcomes associated with nonreportable prenatal cell-free DNA screening results. Am J Obstet Gynecol. 2023 Sep;229(3):300.e1-300.e9. doi: 10.1016/j.ajog.2023.03.026. Epub 2023 Mar 23. PMID 36965866
- [Derived] Dar P, Jacobsson B, MacPherson C, Egbert M, Malone F, Wapner RJ, Roman AS, Khalil A, Faro R, Madankumar R, Edwards L, Haeri S, Silver R, Vohra N, Hyett J, Clunie G, Demko Z, Martin K, Rabinowitz M, Flood K, Carlsson Y, Doulaveris G, Malone C, Hallingstrom M, Klugman S, Clifton R, Kao C, Hakonarson H, Norton ME. Cell-free DNA screening for trisomies 21, 18, and 13 in pregnancies at low and high risk for aneuploidy with genetic confirmation. Am J Obstet Gynecol. 2022 Aug;227(2):259.e1-259.e14. doi: 10.1016/j.ajog.2022.01.019. Epub 2022 Jan 25. PMID 35085538
- [Derived] Dar P, Jacobsson B, Clifton R, Egbert M, Malone F, Wapner RJ, Roman AS, Khalil A, Faro R, Madankumar R, Edwards L, Strong N, Haeri S, Silver R, Vohra N, Hyett J, Demko Z, Martin K, Rabinowitz M, Flood K, Carlsson Y, Doulaveris G, Daly S, Hallingstrom M, MacPherson C, Kao C, Hakonarson H, Norton ME. Cell-free DNA screening for prenatal detection of 22q11.2 deletion syndrome. Am J Obstet Gynecol. 2022 Jul;227(1):79.e1-79.e11. doi: 10.1016/j.ajog.2022.01.002. Epub 2022 Jan 13. PMID 35033576
- See also: 1p36 Deletion Syndrome — http://www.ncbi.nlm.nih.gov/books/NBK1191/
- See also: Angelman Syndrome — http://www.ncbi.nlm.nih.gov/books/NBK1144/
- See also: Cri-du-chat Syndrome — http://www.omim.org/entry/123450?search=number%3A%28123450%29&highlight=123450.